CLINICAL TRIAL: NCT01282359
Title: Efficacy of a Minimal Intervention Educational Program in the Asthma Control and Exacerbations Prevention
Acronym: PROMETEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-PRO-2010-16
Record Dates: First submitted 2011-01-19; First posted 2011-01-25 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: Educational asthma program; Clusters analysis study; Asthma Control Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clinical Practice Group (Other): Patients collected in centres randomized as usual clinical practice, who will not receive the limited educational asthma program.
  Interventions: Other: Clinical practice group
- "Gold Standard" educational group (Other): Patients will receive a formal program of structured and individualized education, enrolled in centres recognized by using high standard procedures in asthma education.
  Interventions: Other: "Gold Standard" educational group
- Intervention group (Other): This group will receive a limited educational asthma program (minimal educational intervention)
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Clinical practice group — Clinical practice group will not receive any specific education
  Arms: Clinical Practice Group
Other: "Gold Standard" educational group — "Gold Standard" educational group will receive a formal program of structured and individualized education
  Arms: "Gold Standard" educational group
Other: Intervention group — Intervention group will take the limited educational asthma program which have three parts: basic information, establishment and revision of a small Action Plan (MiniPlan) and training and review of the inhalation skill of the prescribed device. Educators involved will attend a short workshop (6 h), where they will be trained in the program.
  Arms: Intervention group

SUMMARY:
The asthma clinical practice guidelines categorize with the highest evidence level the effectiveness of educational programs. However, health care professionals not regularly applied it. This may contribute to inadequate control of the disease. Consequently, their designs and implementation strategies should be reviewed.

Hypothesis. An asthma educational program based on a limited intervention, managed by professionals with minimal training in education, could provide a significant decrease in the morbidity of the disease.

Objective. Determine the effectiveness, in terms of prevention of exacerbations (future risk) and improved asthma control (current control) of an educational program based on a reduced or minimal intervention.

DETAILED DESCRIPTION:
Method. A prospective, multicentre, centre randomized ("clusters analysis"), controlled, designed to evaluate the efficacy (reduction of exacerbations) and control degree control (increased ACT score) of an asthma educational program based on a limited intervention in patients with mild to moderate persistent asthma with an ACT <20. The cases included will be distributed into three arms: the intervention group, who will take the limited educational asthma program; clinical practice group, who will not receive any specific education; and education "gold standard" group, which will receive a formal program of structured and individualized education. 250 cases will be including from 25 Spanish centres (pulmonary and primary care): 10 allocated to the intervention group, 10 clinical practice group, and 5 of the gold standard group. Each centre will enrol 10 patients and will be followed for a year in four programmed visits. At baseline and at follow-up visits, will be collected in each patient: ACT score, the number of emergency room visits, unscheduled visits, hospital admissions, cycles of oral prednisone (> 15 days), compliance level, spirometric values and daily dose of inhaled corticosteroid (microg. or equivalent per day). Patients in the intervention group will receive the limited educational asthma program, which have three parts: basic information, establishment and revision of a small Action Plan (MiniPlan) and training and review of the inhalation skill of the prescribed device. Educators involved will attend a short workshop (6 h), where they will be trained in the program.

ELIGIBILITY:
Inclusion Criteria:

* Male and female asthma patients with mild or moderate persistent asthma after treatment according to criteria of the GINA2009.
* Aged 18 and under 70 years.
* With ACT (Asthma Control Test) <20 treated at the outpatient clinics of the participating centers.

Exclusion Criteria:

* Severe exacerbation of asthma (which required emergency room visit and/or hospitalization) within 30 days prior to visit 1.
* Severe disabling comorbidity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations | 1 year
  Patients will be followed for a year in four programmed visits. At baseline and at follow-up visits, will be collected in each patient the number of asthma exacerbations.

SECONDARY OUTCOMES:
ACT score | 1 year
  Patients will be followed for a year in four programmed visits. At baseline and at follow-up visits, will be collected in each patient the Asthma Control Test score.

CONTACTS AND LOCATIONS:
Overall Officials: Antolin Lopez, MD, Study Chair — Hospital Universitario Puerta Hierro Madrid (Spain); Meritxell Peiro, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; José M Ignacio, MD, Study Chair — Hospital Serrania de Ronda. Málaga (Spain).; José A Quintano, MD, Study Chair — Centro de Salud Lucena I. Lucena. Córdoba (Spain).; Santiago Bardagí, MD, Study Chair — Hospital de Mataró. Barcelona (Spain); Vicente Plaza, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Morell F, Genover T, Reyes L, Benaque E, Roger A, Ferrer J. [Monitoring of asthma outpatients after adapting treatment to meet international guidelines]. Arch Bronconeumol. 2007 Jan;43(1):29-35. doi: 10.1016/s1579-2129(07)60017-2. Spanish. PMID 17257561
- [Background] Mansour ME, Rose B, Toole K, Luzader CP, Atherton HD. Pursuing perfection: an asthma quality improvement initiative in school-based health centers with community partners. Public Health Rep. 2008 Nov-Dec;123(6):717-30. doi: 10.1177/003335490812300608. PMID 19711653
- [Background] Henry RL, Gibson PG, Vimpani GV, Francis JL, Hazell J. Randomized controlled trial of a teacher-led asthma education program. Pediatr Pulmonol. 2004 Dec;38(6):434-42. doi: 10.1002/ppul.20095. PMID 15690558